CLINICAL TRIAL: NCT01197456
Title: Predictors of Ovarian Insufficiency Through Serial Exams in Young Breast Cancer Patients (POISE Study)
Brief Title: Predictors of Ovarian Insufficiency in Young Breast Cancer Patients
Acronym: POISE
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: University of Pennsylvania (Other); University of Southern California (Other); American Cancer Society, Inc. (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor of Obstetrics, Gynecology, and Reproductive Sciences, University of California, San Diego
Other Study IDs: UCSD POISE; K23HD058799 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Ovarian Insufficiency; Ovarian Failure
Keywords: Breast cancer; Ovarian insufficiency; Ovarian failure; Reproduction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed/chemotherapy: Breast cancer patients who will undergo chemotherapy
- Unexposed: Breast cancer patients who will not undergo chemotherapy

SUMMARY:
More than two million American women are breast cancer survivors. Approximately one-third of these women are premenopausal at diagnosis and face issues related to reproduction as they undergo cancer treatment. Ovarian function after breast cancer diagnosis has implications on breast cancer prognosis, choice of adjuvant therapy and reproductive issues such as desire for fertility or concerns about menopause. Therefore, tools to accurately predict ovarian function in breast cancer survivors could significantly impact physicians and patients in counseling, medical and surgical treatment choices, and consideration of fertility preservation options.

The goal of this proposal is to identify pre-chemotherapy hormonal, genetic and ovarian imaging markers that can predict ovarian failure and characterize the course of ovarian function after chemotherapy. The investigators plan to follow a group of young women from breast cancer diagnosis to five years after chemotherapy. The investigators will study the following risk factors: blood hormone levels that reflect ovarian function, genetic mutations that affect how individuals metabolize chemotherapy, and ovarian size and egg count by MRI and ultrasound. The investigators hypothesize that these biomarkers are related to risk of ovarian insufficiency singly. After examining these individual risk factors for ovarian failure, the investigators will put them together into an Ovarian Failure Clinical Predictive Index. This index will be a tool similar to the Gail Model that can be used to determine individual risk for ovarian failure. This tool would assist young breast cancer patients and their physicians in making treatment decisions that would impact cancer survival and reproduction.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of breast cancer (Stages 0-III)
* Age <=45
* Premenopausal (at least one menses over past year)
* Has a uterus and at least one ovary

Exclusion Criteria:

* Prior chemotherapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Newly diagnosed breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Su HC, Haunschild C, Chung K, Komrokian S, Boles S, Sammel MD, DeMichele A. Prechemotherapy antimullerian hormone, age, and body size predict timing of return of ovarian function in young breast cancer patients. Cancer. 2014 Dec 1;120(23):3691-8. doi: 10.1002/cncr.28942. Epub 2014 Jul 31. PMID 25081546
- [Result] Homer MV, Charo LM, Natarajan L, Haunschild C, Chung K, Mao JJ, DeMichele AM, Su HI. Genetic variants of age at menopause are not related to timing of ovarian failure in breast cancer survivors. Menopause. 2017 Jun;24(6):663-668. doi: 10.1097/GME.0000000000000817. PMID 28118297
- [Result] Su HI, Sammel MD, Homer MV, Bui K, Haunschild C, Stanczyk FZ. Comparability of antimullerian hormone levels among commercially available immunoassays. Fertil Steril. 2014 Jun;101(6):1766-72.e1. doi: 10.1016/j.fertnstert.2014.02.046. Epub 2014 Apr 14. PMID 24726216

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exposed/Chemotherapy | Unexposed
Started | 171 | 61
Completed | 171 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed/Chemotherapy | Unexposed | Total
Number analyzed (Participants) | 171 | 61 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 171 | 61 | 232
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (5.1) | 41.0 (5.7) | 39.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 61 | 232
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 171 | 61 | 232

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Ovarian Insufficiency (Without of Menses for 12 Months) After Breast Cancer Diagnosis
Description: Number of participant without of menses for 12 months after breast cancer diagnosis
Time Frame: Years 1-5
Population: 25 participants could not be evaluated for this outcome due to censoring for cancer recurrence, death, bilateral salpingo-oophorectomy, or hysterectomy.
  38 additional participants could not be evaluated for this outcome due to loss to follow up.
Measure: Number; unit: Participants
Arm/Group | Exposed/Chemotherapy | Unexposed
Number analyzed (Participants) | 128 | 41
Participants | 27 | 11

2. Secondary Outcome: Number of Participants Who Experience Return of Menses After 3 Months of Amenorrhea
Description: Number of participants who experience return of menses after 3 months of amenorrhea
Time Frame: Years 1-5
Population: We did not undertake this analysis for participants who did not undergo chemotherapy (unexposed) or were censored for recurrence, death, hysterectomy or bilateral salpingo-oophorectomy (n=108) as this measure is not applicable
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed/Chemotherapy | Unexposed
Number analyzed (Participants) | 124 | 0
Participants | 62 | 0

ADVERSE EVENTS:
Arm/Group | Exposed/Chemotherapy | Unexposed
All-Cause Mortality (participants affected / at risk) | 2/171 | 1/61
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/61
Other Adverse Events (participants affected / at risk) | 0/171 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No